CLINICAL TRIAL: NCT05032820
Title: Phase II Multicenter Trial of Anti-BCMA CAR T-Cell Therapy for MM Patients With Sub-Optimal Response After Auto HCT and Maintenance Len. BMTCTN1902
Brief Title: Upfront Chimeric Antigen Receptor T-Cell to Upgrade Response in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marcelo Pasquini, MD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other); Celgene a wholly owned subsidiary of BMS (Unknown)
Responsible Party: Sponsor-Investigator, Marcelo Pasquini, MD, Primary Investigator, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN1902; 2U10HL069294-11 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2021-07-08; First posted 2021-09-02 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; CAR T-cells; Anti-Myeloma Agents; lenalidomide; Maintenance Therapy; Hematologic Disorders; Infusion
MeSH Terms: conditions — Multiple Myeloma; Hematologic Diseases | interventions — Lenalidomide; idecabtagene vicleucel; Cyclophosphamide; fludarabine; Leukapheresis

STUDY DESIGN:
Intervention Model Description: Assess anti-B Cell Maturation Antigen(BCMA) chimeric antigen receptor (CAR) T-cells (bb2121) to improve post autologous hematopoietic cell transplant (HCT) responses among patients with multiple myeloma (MM).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide and bb2121 (Experimental): Patients complete apheresis and proceed to lymphodepleting chemotherapy with cyclophosphamide 300mg/m^2 and fludarabine 30mg/m^2 for 3 consecutive days followed by the infusion of BCMA CAR T-cells at a target dose of 450 x10^6 cells. Maintenance lenalidomide, starting at 5mg a day for 21 days of a 28-day cycle will be initiated at a minimum of at least 30 days, but no later than 180 days after the CAR T-cell infusion and will continue until the patient reaches 12 months post CAR T-cell infusion and continue free of progression.
  Interventions: Drug: Lenalidomide; Biological: bb2121; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: leukapheresis

INTERVENTIONS:
Drug: Lenalidomide — Maintenance lenalidomide, starting at 5 mg a day for 21 days of a 28-day cycle, will be initiated at a minimum of at least 30 days, but no later than 180 days after the CAR T-cell infusion and will continue until the participant reaches 12 months post CAR T-cell infusion and continues free of progression
  Other Names: Revlimid
Biological: bb2121 — Participants receive infusion of BCMA CAR T-cells at a target dose of 450 x 10^6 cells.
  Other Names: ide-cel
Drug: Cyclophosphamide — 300 mg/m^2/day for 3 consecutive days prior to the CAR T infusion
Drug: Fludarabine — 30 mg/m^2/day or 3 consecutive days prior to the CAR T infusion
Procedure: leukapheresis — Placement of central line catheter and leukapheresis

SUMMARY:
This study is designed as a Phase II, multicenter, single arm trial to assess anti-B Cell Maturation Antigen (BCMA) chimeric antigen receptor (CAR) T-cells (bb2121) to improve post autologous hematopoietic cell transplant (HCT) responses among patients with multiple myeloma (MM).

DETAILED DESCRIPTION:
After meeting the eligibility criteria and enrolling on the trial, patients will undergo leukapheresis for collection of autologous lymphocytes, which will be sent to BMS/Celgene manufacturing facilities. Once cells have been manufactured, patients will then proceed to lymphodepleting chemotherapy with cyclophosphamide 300mg/m^2 and fludarabine 30mg/m^2 for 3 consecutive days followed by the infusion of BCMA CAR T-cells at a target dose of 450 x10^6 cells. Maintenance lenalidomide, starting at 5mg a day for 21 days of a 28-day cycle will be initiated at a minimum of at least 30 days, but no later than 180 days after the CAR T-cell infusion and will continue until the patient reaches 12 months post CAR T-cell infusion and continue free of progression

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18.00 years
2. Patients must meet the criteria for symptomatic MM requiring therapy (Appendix A) prior to initiating initial systemic anti-myeloma treatment.
3. Patients must have received initial systemic anti- myeloma therapy consisting of induction therapy and consolidation with high-dose melphalan (>140 mg/m^2 ) followed by an auto HCT (minimum cell dose of 2x10^6 CD34+ cells/kg (actual body weight) within 12 months from initiation of systemic anti-myeloma therapy.
4. Patient must have additional stored stem cells greater than or equal to 2x10^6 CD34+ cells per kg actual body weight.
5. Patients must be less than or equal to 12 months after autologous HCT at the time of enrollment.
6. Patients must have initiated maintenance therapy with lenalidomide-based regimen within 6 months after the auto HCT and have received at least 3 months of maintenance prior to enrollment.
7. Patients must have tolerated a minimum dose of lenalidomide 5 mg/day for 21 days of a 28-day cycle for greater than 2 cycles without having to stop due to toxicities.
8. Patients must have a VGPR or less (Section 3.1) in reference to time time of initiation of initial systemic anti-myeloma therapy at study enrollment.
9. Patients must have Karnofsky performance greater than or equal to 70.
10. Patients must have recovered to Grade 1 or baseline of any non-hematologic toxicities due to prior treatments, excluding Grade 2 neuropathy.
11. Absolute neutrophil count (ANC) greater than or equal to 1,500/mm3 without filgrastim use in the prior 14 days.
12. Platelet count greater than 100,000/mm^3 (without platelet transfusion in the previous 7 days or thrombopoietin mimetics in the previous 28 days).
13. Hemoglobin greater than 9 g/dL (without red blood cell transfusion in the previous 7 days).
14. Creatinine Clearance (CrCl) greater than or equal to 60 mL/min, measured or estimated by Cockcroft-Gault equation.
15. Corrected serum calcium less than or equal to 13.5 mg/dL.
16. Oxygen saturation greater than 92% on room air.
17. Hepatic Function: a. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x upper limit of normal (ULN) b. Serum total bilirubin less than or equal to 2 x ULN. Patients who have been diagnosed with Gilbert's disease are permitted to exceed the defined bilirubin value of 2 x ULN
18. International ratio (INR) or partial thromboplastin time (PTT) less than 1.5 x ULN
19. Cardiac Function: left ventricular ejection fraction greater than 45% by echocardiogram or MUGA.
20. Patients must be willing and able to adhere to the study visit schedule and other protocol requirements including regulatory requirement of a 15 year follow up using the CIBMTR long term follow up mechanism.
21. Female patients of childbearing potential (FCBP1 ) must: a. Have a negative serum pregnancy test with a sensitivity of at least 50 mIU/mL prior to enrollment b. Agree to use, and be able to comply with, TWO acceptable methods of birth control (Appendix C), one highly effective method and one additional effective (barrier) method AT THE SAME TIME, from screening through at least 1 year following bb2121 infusion or 4 weeks following discontinuation of lenalidomide, whichever is later. c. Agree to abstain from breastfeeding from screening through at least 1 year following bb2121 infusion or 4 weeks following discontinuation of lenalidomide, whichever is later.
22. Male patients must: a. Agree to use a condom during sexual contact with a pregnant female or a FCBP, even if he has undergone a successful vasectomy, from screening through at least 1 year following bb2121 infusion or 4 weeks following discontinuation of lenalidomide whichever is later b. Must not donate sperm from screening through at least 1 year following bb2121 infusion or 4 weeks following discontinuation of lenalidomide whichever is later.

Exclusion Criteria:

1. Patients with a prior allogeneic hematopoietic cell.
2. Female of childbearing potential (FCBP) is a female who:

   * has achieved menarche at some point,
   * has not undergone a hysterectomy or bilateral oophorectomy or
   * has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
3. Patients with disease progression (see Section 3.1.2 for disease progression definition) at any time prior to enrollment.
4. Patients receiving any of the following less than 14 days prior to enrollment:

   1. Plasmapheresis
   2. Major surgery (as defined by the investigator)
   3. Radiation therapy other than local therapy for MM-associated bone lesions
   4. Use of any systemic anti-myeloma drug therapy (with the exception of lenalidomide maintenance)
   5. Any investigational agents
   6. Corticosteroids (Physiologic replacement, topical, intranasal and inhaled steroids are permitted)
5. Patients with known Central Nervous System (CNS) involvement with MM.
6. Patients with a prior organ transplant requiring systemic immunosuppressive therapy.
7. Patients who previously experienced toxicities related to lenalidomide resulting in permanent treatment discontinuation.
8. Patients who experienced thromboembolic events while on full anticoagulation during prior therapy with an immunomodulatory agent (IMiD).
9. Patients unwilling to take DVT prophylaxis while on lenalidomide maintenance.
10. Patients with history of greater than or equal to Grade 2 hemorrhage within 30 days of enrollment.
11. Patient requiring ongoing treatment with chronic, therapeutic dosing of anticoagulants (e.g. Warfarin, low molecular weight heparin, Factor Xa inhibitors).
12. Patients with history or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, subarachnoid hemorrhage or other CNS bleed, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
13. Patients with active or history of plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or clinically significant amyloidosis.
14. Patients with purely non-secretory MM [prior to starting systemic therapy, absence of a monoclonal protein (M protein) in serum as measured by electrophoresis and immunofixation and the absence of Bence Jones protein in the urine defined by use of conventional electrophoresis and immunofixation techniques and the absence of involved serum free light chain greater than 100mg/L]. Patients with light chain MM detected in the serum by free light chain assay are eligible.
15. Patients with a history of Class III or IV congestive heart failure (CHF) or severe nonischemic cardiomyopathy, unstable or poorly controlled angina, myocardial infarction, or hemodynamically significant ventricular arrhythmia within the previous 6 months prior to starting study treatment.
16. Patients with ongoing treatment with chronic immunosuppressants (e.g. cyclosporine or systemic steroids at any dose). Physiologic replacement, intermittent topical, inhaled or intranasal corticosteroids are allowed.
17. Patients with active clinically significant autoimmune disease, defined as a history of requiring systemic immunosuppressive therapy and at ongoing risk for potential disease exacerbation. Patients with a history of autoimmune thyroid disease, asthma, or limited skin manifestations are potentially eligible.
18. Patients seropositive for human immunodeficiency virus (HIV-1), chronic or active hepatitis B or C, or acute hepatitis A. If any history of exposure to hepatitis B or C then DNA PCR should be negative.
19. Patients with previous history of treatment with any gene therapy-based therapeutic for cancer or investigational cellular therapy for cancer or BCMA targeted therapy.
20. Patients with prior malignancies except resected basal cell carcinoma or treated carcinoma in situ. Cancer treated with curative intent less than 5 years prior to enrollment will not be allowed unless approved by the Protocol Officer or one of the Protocol Chairs. Cancer treated with curative intent greater than 5 years prior to enrollment is allowed.
21. Female patients who are pregnant (positive beta-HCG), or breastfeeding, or who intend to become pregnant during participation in the study.
22. Patient with known allergy or hypersensitivity to any of the study medications, their analogues, or excipients in the various formulations of any agent.
23. Patient with serious medical of psychiatric illness likely to interfere with participation on this clinical study.
24. Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment.
25. Patients unwilling or unable to provide informed consent 25. Patients unable or unwilling to return to the transplant center for treatment and follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2025-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo C Pasquini, MD, MS, Study Director — Medical College of Wisconsin; Alfred Garfall, MD, Principal Investigator — University of Pennsylvannia; Sergio Giralt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (15):
- United States (15):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Roswell Park Cancer Center, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania Hospital Center, Philadelphia, Pennsylvania
  - Baylor College and Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc., where indicated).
Supporting Information: Study Protocol
Time Frame: Within 6 months of official study closure at participating sites
Access Criteria: Available to public
URL: https://biolincc.nhlbi.nih.gov/home

REFERENCES:
- See also: Blood and Marrow Transplant Clinical Trials Network Website — https://bmtctn.net/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: BMT CTN 1902's enrollment was between January 2022 and December 2023 with 40 participants enrolled from 12 centers. The study opened to accrual in February 2021. Fifteen centers were activated for enrollment. The study closed to accrual on January 09, 2024.
Pre-assignment Details: There was a Safety Run-in that included the first three participants enrolled on the study with staggered enrollment to assess for excess early toxicity. These data were reviewed and enrollment was approved in the Continuing Enrollment Phase which began on October 14, 2022.
Period: Overall Study
Arm/Group | Lenalidomide and bb2121
Started | 40
Completed | 38
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Enrolled Participants
Arm/Group | Lenalidomide and bb2121
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Infusion (years) Population: This row is only for infused patients and therefore has less participants in this row than others as not all enrolled participants were infused.
  years
    number analyzed (Participants) | 38
    (all) | 61.2 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 29
  More than one race | 1
  Unknown or Not Reported | 3
Karnofsky Performance Score [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead
  Participants
    70 or 80 | 17
    90 or 100 | 23
Multiple Myeloma Paraprotein Type [Count of Participants; unit: Participants] — There are 5 types of heavy chains: IgG, IgA, IgD, IgE, and IgM. There are 2 types of light chains: kappa and lambda Immunoglobulins are made up of a heavy chain and a light chain. The diagnosis of myeloma is labelled according to the type of immunoglobulin that has become abnormal.
  Participants
    IgA Kappa | 2
    IgA Lambda | 2
    IgG Kappa | 20
    IgG Lamda | 6
    Kappa light chain | 8
    Lambda light chain | 2
ISS Stage at Diagnosis [Count of Participants; unit: Participants] — Stage I: Serum B2 microglobulin < 3.5mg/L; serum albumin >= 3.5 g/dL Stage II: Serum B2 microglobulin < 3.5mg/L; serum albumin < 3.5 g/dL; OR Serum B2 microglobulin 3.5 to 5.5 mg/L, irrespective of serum albumin Stage III: Serum B2 microglobulin > 5.5. mg/L
  Participants
    I | 14
    II | 18
    III | 6
    Unknown | 2
R-ISS Stage at Diagnosis [Count of Participants; unit: Participants] — Stage I: Serum B2 microglobulin < 3.5 mg/L; Serum albumin >= 3.5 g/dL; Standard-risk chromosomal abnormalities (CA) by iFISH; normal lactate dehydrogenase levels (LDH) Stage II: Nor R-ISS Stage I or III Stage III: Serum B2 microglobulin >= 5.5 mg/L and either high risk CA by iFISH or high LDH
  Participants
    I | 11
    II | 20
    III | 2
    Unknown | 7
Cytogenetics [Count of Participants; unit: Participants] — Cytogenetic abnormalities can assess the risk and prognosis of multiple myeloma. High risk includes t(4;14), t(14;16), t(14;20), del17p, 1q amplification, and >=2 HRCA. Standard risk includes chromosomal hyperdiploid. High risk indicates worse outcomes.
  Participants
    High risk | 9
    No abnormalities | 7
    Standard risk | 23
    Unknown | 1
Myeloma Risk Status [Count of Participants; unit: Participants] — myeloma risk defines high risk disease based on ISS 3 and or high risk cytogenetics (t(4;14), t(14;16), t(14;20), deletion 17p or p53 deletion or amplification of 1q). Others are included in standard risk. High risk indicates worse outcomes.
  Participants
    High risk | 12
    Standard risk | 28
Number of Lines of Initial Systemic Anti-Myeloma Therapy [Count of Participants; unit: Participants]
  1 Line | 32
  2 Lines | 6
  3 Lines | 2
Disease Status Prior to Transplant [Count of Participants; unit: Participants] — PR: >=50% reduction (RED) in serum monoclonal paraprotein (PP) & RED in 24hr urinary monoclonal PP by >=90% or to <200 mg/24hr; or if M protein unmeasurable: >=50% RED in difference b/w involved & uninvolved FLC levels or 50% RED of involved FLC w/ 50% RED in ratio; or only bone marrow (BM) measurable: >=50% RED in BM plasma cells if baseline >=30%; or >=50% RED in size of soft tissue plasmacytomas. VGPR: PR & Serum or urine PP detectable by immunofixation but not electrophoresis; OR >=90% serum PP RED + urine PP <100 mg/24hr & >90% involved light chain RED. SD: none of above & no progression.
  Participants
    VGPR | 7
    PR | 30
    SD | 3
Disease Status Prior to Enrollment [Count of Participants; unit: Participants] — MR: >=25% & <50% RED in serum monoclonal PP and RED in 24hr urinary monoclonal protein by 50-89%; or >=50% RED in size of soft tissue plasmacytomas if present at baseline.
  Participants
    VGPR | 22
    PR | 17
    MR | 1
Disease Status at LD Chemotherapy Initiation [Count of Participants; unit: Participants]
  VGPR | 22
  PR | 13
  MR | 1
  Missing | 2
  No LD Chemotherapy | 2
Interval from Diagnosis of Symptomatic Multiple Myeloma to Transplant [Mean (Standard Deviation); unit: months] — Interval is calculated as (Date of transplant - date of diagnosis of symptomatic multiple myeloma +1)/(365.25/12)
  months | 7.1 (2.34)
interval from diagnosis of symptomatic Multiple Myeloma to enrollment [Mean (Standard Deviation); unit: months] — Interval is calculated as (Date of enrollment - date of diagnosis of symptomatic multiple myeloma +1)/(365.25/12)
  months | 16.2 (2.77)
Interval from Transplant to Enrollment [Mean (Standard Deviation); unit: months] — Interval is calculated as (Date of enrollment - date of transplant +1)/(365.25/12)
  months | 9.1 (1.68)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of BCMA CAR-T Cell Therapy
Description: Achieving a complete response or better (CR or sCR) as assessed by the 6-month time point after BCMA CAR T-cell therapy in MM patients with suboptimal disease responses after an autologous HCT and lenalidomide maintenance.
Time Frame: 6 months
Population: Patients who received BCMA CAR T-Cell Therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide and bb2121
Number analyzed (Participants) | 38
Participants
  Acheived CR/sCR by 6 Months post Infusion | 25
  Did Not Acheive CR/sCR by 6 Months post Infusion | 13
Statistical Analysis 1: Comparison: Lenalidomide and bb2121; Test type: Superiority; p < 0.0001, Fisher Exact — p-value is calculated using Fisher's exact test and is a one-sided test with a 5% significance level that tests whether the proportion of successes is greater than 10%; One-sided test with a 5% significance level that tests whether the proportion of successes is greater than 10%; Proportion of Patients Achieving CR/sCR = 65.8, 90% CI 2-sided [51.2 to 78.4]

2. Secondary Outcome: Assessment of Disease Progression
Description: Diseases will be assessed by response categories based on the International Myeloma Working Group: Stringent Complete Response (sCR), Complete Remission (CR), Very Good Partial Remission (VGPR), Partial Remission (PR), Minimal Response (MR), Stable Disease (SD).
Time Frame: 1 Year
Reporting Status: Not Posted

3. Secondary Outcome: Best Disease Response
Description: : Proportion of patients achieving upgrade in response following enrollment (SD to MR or greater, MR to PR or greater, or PR to VGPR or greater) and Conversion to MRD negativity. MRD will be assessed by multi-color flow at 10-5 level
Time Frame: 1 Year
Reporting Status: Not Posted

4. Secondary Outcome: Non Relapse Mortality
Description: Non-Relapse Mortality (NRM) is defined as death occurring in a patient from causes other than disease relapse or progression. Disease progression is the competing event for NRM.
Time Frame: 1 Year
Reporting Status: Not Posted

5. Secondary Outcome: Progression Free Survival
Description: Defined as progression of disease or death from any cause. Surviving patients without disease progression will be censored at the date of last contact.
Time Frame: 1 Year
Reporting Status: Not Posted

6. Secondary Outcome: Incidence of Cytokine Release Syndrome
Description: Overall incidence of CRS of any grade and grade 3 or 4 CRS post CAR T-cell infusion will be reported on all patients.
Time Frame: 1 year
Reporting Status: Not Posted

7. Secondary Outcome: Incidence of Prolonged Cytopenias
Description: Overall incidence of prolonged cytopenias will be reported. Prolonged cytopenia is defined as failure to achieve ANC greater than 500/mm3 or platelet count greater than 20,000/mm3(with or without support) by 30 days post CAR T-cell ifusion.
Time Frame: 1 Year
Reporting Status: Not Posted

8. Secondary Outcome: Incidence of Neurotoxicity
Description: Overall incidence of CAR T-cell related neurotoxicity per the ASBMT immune effector cell associated neurotoxicity syndrome (ICANS) Consesus Grading.
Time Frame: 1 Year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Exploratory Objective 1: Incidence of Toxicities Greater Than or Equal to Grade 3 Per the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: All Grade 3 or higher toxicities will be tabulated. The proportion of patients experiencing cytokine release syndrome CRS will be reported including overall and grades 3-4 based on the ASTCT grading
Time Frame: 1 Year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory Objective 2: Incidence of Infections Per Protocol-specific Manual of Procedures (MOP)
Description: incidence of definite and probable viral, fungal and bacterial infections will be tabulated for each patient
Time Frame: 1 Year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Exploratory Objective 3: Maintenance Feasibility
Description: The feasibility of resuming maintenance following enrollment by 180 days after CAR T-cell infusion will be described. The proportion of patients initiating maintenance at 180 days following bb2121 infusion will be reported.
Time Frame: 1 Year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Exploratory Objective 2: Overall Survival
Description: The event is death from any cause. The time to this event is the time from initial enrollment to sdeath, loss to follow-up, or the end of the study, whichever comes first.
Time Frame: 1 Year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Exploratory Objective 2: CAR Tcell Expansion
Description: Quantitation of CAR T-cells in peripheral blood will be determined at specified timepoints by quantitative PCR assay, measured in copies/mcg genomic DNA. Peak CAR T-cell expansion will be compared between subjects who are and are not in CR at 12 months, and between subjects who are and are not progression-free at 12 months.
Time Frame: 1 Year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Exploratory Objective 2: CAR T-cell Persistence
Description: Quantitation of CAR T-cells in peripheral blood will be determined at specified timepoints by quantitative PCR assay, measured in copies/mcg genomic DNA. Persistence will be measured in 2 ways: 1) as an area under the curve (AUC) over first 6 months post CAR T-cell infusion; and 2) as still having detectable CAR T-cells at 6 months post CAR T-cell infusion. AUC6mos and 6- month persistence will be compared between subjects who are and are not in CR at 12 months, and between subjects who are and are not progression-free at 12 months.
Time Frame: 1 Year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Exploratory Objective 2: BCMA Expression
Description: BCMA expression at specified timepoints will be determined by immunohistochemical staining of bone marrow biopsy specimens and/or flow cytometric analysis of bone marrow aspirate material, in order to assess for baseline expression and potential loss of expression post-treatment. Both percent of MM cells that stain positive as well as staining intensity will be reported.
Time Frame: 1 Year
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Exploratory Objective 2: Immune Reconstitution
Description: The cellular composition of marrow (T-Cells, B-Cells, Natural Killer Cells, dendritic cells, and myeloid derived suppressor cells) will be quantified at the specified timepoints by flow cytometry.
Time Frame: 1 Year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All SAEs and AEs were collected from enrollment to study completion, or for 12 months after bb2121 infusion.
Description: Adverse events are collected on the adverse event form, toxicity form, and myelotoxicity form.
Arm/Group | Lenalidomide and bb2121
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 9/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and bb2121 (N=40)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Cytokine Release Syndrome (Immune system disorders) | 5 (5)
Pneumonia (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and bb2121 (N=40)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood alkaline phosphatase (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (9)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Embolism (Vascular disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count decreased (Investigations) | 34 (129)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophil count decreased (Investigations) | 31 (98)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 3 (6)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (3)
Sinusitis (Infections and infestations) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 29 (65)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2)
Paraesthesia (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Oedema (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT05032820/Prot_003.pdf
  • Statistical Analysis Plan (2025-08-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT05032820/SAP_004.pdf
  • Informed Consent Form: Informed Consent to Participate in Research (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT05032820/ICF_001.pdf
  • Informed Consent Form: Pregnancy Partner Informed Consent Form (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT05032820/ICF_002.pdf